CLINICAL TRIAL: NCT05646836
Title: A Phase Ib, Open-label, Multicenter Dose-escalation Study to Evaluate the Safety, Pharmacokinetics, and Activity of XmAb24306 in Combination With Cevostamab in Patients With Relapsed/Refractory Multiple Myeloma
Brief Title: A Study to Evaluate the Safety, Pharmacokinetics, and Activity of XmAb24306 in Combination With Cevostamab in Participants With Relapsed/Refractory Multiple Myeloma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GO43980; 2022-001204-18 (EudraCT Number); 2023-505212-38-00 (Other: EU CT Number)
Record Dates: First submitted 2022-12-02; First posted 2022-12-12 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — tocilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: Dose-Escalation and Expansion: XmAb24306+Cevostamab (Experimental): Participants will receive escalating doses of XmAb24306 with a fixed dose regimen for cevostamab up to the maximum tolerated dose (MTD). After dose escalation has been completed, up to two expansion cohorts each investigating different XmAb24306 doses in combination with cevostamab may be enrolled.
  Interventions: Drug: Cevostamab; Drug: XmAb24306; Drug: Tocilizumab
- Arm B: Single-Agent Cevostamab Expansion (Experimental): Participants will receive cevostamab alone.
  Interventions: Drug: Cevostamab; Drug: Tocilizumab

INTERVENTIONS:
Drug: Cevostamab — Cevostamab will be administered intravenously on a 28-day cycle, for up to one year of treatment depending on clinical response.
  Other Names: RO7187797
Drug: XmAb24306 — XmAb24306 will be administered intravenously on a 28-day cycle, for up to one year of treatment depending on clinical response.
  Other Names: RO7310729
  Arms: Arm A: Dose-Escalation and Expansion: XmAb24306+Cevostamab
Drug: Tocilizumab — Tocilizumab will be administered for the treatment of cytokine release syndrome (CRS) when necessary.
  Other Names: Actemra, RoActemra

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics, and activity of XmAb24306 in combination with cevostamab in participants with relapsed/refractory multiple myeloma (R/R MM) who have received a minimum of three prior treatments, including at least one immunomodulatory drug (IMiD), one proteasome inhibitor (PI), and one anti-CD38 monoclonal antibody.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Life expectancy of at least 12 weeks
* Participants must have received a minimum of 3 prior lines of therapy, including at least one PI, one IMiD, and an anti-CD38 monoclonal antibody.
* Documented evidence of progressive disease on or after the last prior therapy, or participants who were intolerant to the last prior therapy.
* Measurable disease, as defined by the protocol
* Participants agree to follow contraception or abstinence requirements as defined in the protocol

Exclusion Criteria:

* Any anti-cancer therapy within 3 weeks prior to initiation of study treatment with exception defined by the protocol
* Participants with autologous stem cell transplantation (SCT) within 100 days prior to first dose of study treatment
* Participants with prior allogeneic SCT or solid organ transplantation
* Known history of hemophagocytic lymphohistiocytosis (HLH) or macrophage activation syndrome (MAS)
* Active or history of autoimmune disease
* Participants with current or history of Central Nervous System (CNS) disease, or current CNS involvement by Multiple Myeloma (MM)
* Significant cardiovascular disease
* Participants with known clinically significant liver disease
* Symptomatic active pulmonary disease requiring supplemental oxygen
* Known active infection requiring intravenous anti-microbial therapy within 14 days prior to first study drug administration
* Any episode of active, symptomatic COVID-19 infection, or requiring treatment with IV antivirals for COVID-19 (not including COVID-19 primary prophylaxis) within 14 days, prior to first study treatment
* Other protocol defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-03-21 (Actual); Primary Completion 2026-11-18 (Estimated); Study Completion 2026-11-18 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with Adverse Events (AEs) | Up to approximately 3 years
  Adverse events will be reported according to the National Cancer Institute Common Terminology Criteria for Adverse Events, Version 5.0 (NCI CTCAE v5.0), and Cytokine Release Syndrome (CRS), will be graded based on the American Society for Transplantation and Cellular Therapy (ASTCT) criteria.

SECONDARY OUTCOMES:
Serum Concentration of XmAb24306 | Up to approximately 3 years
Serum Concentration of Cevostamab | Up to approximately 3 years
Objective Response Rate (ORR) | Up to approximately 3 years
  ORR will be determined by the investigator according to International Myeloma Working Group (IMWG) criteria.
Rate of Complete Response (CR)/ Stringent Complete Response (sCR) | Up to approximately 3 years
  Rate of CR/sCR will be determined by the investigator.
Rate of Very Good Partial Response (VGPR) | Up to approximately 3 years
  Rate of VGPR will be determined by the investigator.
Percentage of Participants With Anti-Drug Antibodies (ADA) to XmAb24306 and Cevostamab | Up to approximately 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (13):
- Australia (3):
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Peter Maccallum Cancer Centre, Melbourne, Victoria
  - Alfred Hospital, Melbourne, Victoria
- Sygehus Lillebaelt - Vejle Sygehus, Vejle, Denmark
- Greece (2):
  - Evangelismos General Hospital of Athens, Athens
  - University of Athens, Hematological Clinic,, Athens
- Israel (2):
  - Rabin Medical Center-Beilinson Campus, Petah Tikva
  - Tel Aviv Sourasky Medical Center PPDS, Tel Aviv
- Oslo University Hospital Rikshospitalet, Oslo, Norway
- South Korea (2):
  - Severance Hospital, Yonsei University, Seoul
  - Asan Medical Center - PPDS, Seoul
- Spain (2):
  - Clinica Universidad de Navarra, Pamplona, Navarre
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing